CLINICAL TRIAL: NCT07171814
Title: Cohort Study of Honghua Xiaoyao Tablet in the Treatment of Premenstrual Syndrome Based on Target Trial Emulation Framework
Brief Title: Cohort Study of Honghua Xiaoyao Tablets in the Treatment of Premenstrual Syndrome Based on Target Trial Emulation Framework
Acronym: TTE
Status: Not yet recruiting | Type: Observational
Sponsor: Lianxin Wang (Other)
Collaborators: Chaoyangmen Community Health Service Center of Dongcheng District in Beijing (Unknown); Hepingli Community Health Service Center,Dongcheng District,Beijing (Unknown)
Responsible Party: Sponsor-Investigator, Lianxin Wang, Principal Investigator, China Academy of Chinese Medical Sciences
Organization: China Academy of Chinese Medical Sciences (Other)
Other Study IDs: Honghua Xiaoyao Tablets; 2022YFC3502004 (Other Grant/Funding Number: National Key R&D Program of China)
Record Dates: First submitted 2025-09-06; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Premenstrual Syndrome
Keywords: Honghua Xiaoyao tablet; Target trial emulation; The real world
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Honghua Xiaoyao tablets: The intervention for this cohort includes treatment with Honghua Xiaoyao Tablets.
  Interventions: Drug: Honghua Xiaoyao tablets

INTERVENTIONS:
Drug: Honghua Xiaoyao tablets — The non-exposed group (patients who did not receive Honghua Xiaoyao Tablets or other targeted drug treatments) only received routine clinical observation, and no drug intervention was applied after obtaining informed consent. If patients need to withdraw from the study due to their condition during the study period, on the premise that the patients have given full informed consent, doctors shall recommend other treatment regimens in accordance with clinical standards (when necessary, first-line drugs such as selective serotonin reuptake inhibitors (SSRIs) may be selected for intervention).
  Other Names: serotonin reuptake inhibitors (SSRIs)

SUMMARY:
To evaluate the efficacy and safety of Honghua Xiaoyao tablets in the treatment of premenstrual syndrome, and the results were further analyzed and evaluated by target trial simulation (TTE) framework.

DETAILED DESCRIPTION:
In this study, the patients in the exposed group were treated with Honghua Xiaoyao Tablets, which were provided by Jiangxi Puzheng Pharmaceutical Co., Ltd. The administration method of this drug was oral: 4 tablets each time, 3 times a day, for a continuous medication period of 3 months. Doctors were required to provide detailed guidance on medication use and record prescriptions; during follow-up visits, the remaining drugs should be checked to track patients' medication adherence.

The patients in the non-exposed group did not use Honghua Xiaoyao Tablets or other targeted drugs, and only received routine clinical observation. No drug intervention was applied to them after obtaining informed consent. However, they completed the follow-up plan as well as various efficacy and safety assessments simultaneously with the exposed group. If patients needed to withdraw from the study due to their condition during the study period (in accordance with the Management of Premenstrual Disorders: ACOG Clinical Practice Guideline No. 7, this applied when premenstrual dysphoric disorder (PMDD) or premenstrual syndrome (PMS) symptoms occurred during follow-up and the patient could not tolerate them), on the premise that the patient had given full informed consent, doctors could recommend first-line drugs such as selective serotonin reuptake inhibitors (SSRIs) for intervention and other treatment regimens in accordance with clinical standards. At the same time, the reasons for the patient's withdrawal and subsequent treatment status should be recorded in detail.

Time zero was defined as the start of the treatment period, i.e., when the doctor issued the prescription. Follow-up visits began at this point, with one follow-up visit conducted every month. The follow-up period covered the 3-month medication period and 1 month after drug discontinuation. This clinical observational study was scheduled to be completed within 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-40 years old (both ends included);
2. According to the 8th edition of "Obstetrics and Gynecology" (2014), patients diagnosed with premenstrual syndrome;
3. In accordance with the TCM syndrome differentiation standard of liver depression and qi stagnation.

Exclusion Criteria:

1. those who were allergic to the ingredients and excipients of Honghua Xiaoyao tablet (exposure group);
2. In the non-exposed group, those receiving or planning to receive other targeted medications for PMS, such as serotonin reuptake inhibitors (SSRIs), hormones, etc.;
3. irregular menstrual cycle (menstrual cycle not within 28±7 days);
4. serious diseases of cardiovascular, cerebrovascular, hematopoietic system, liver and kidney, and malignant tumors;
5. pregnant or lactating women, or those who plan to become pregnant within 6 months;
6. patients with mental illness and alcohol or drug dependence; Patients with other complicated lesions were not eligible for this study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The somatic symptoms included headache, abdominal distension, limb swelling, breast pain, and insufficient motor coordination. Mental symptoms included irritability, emotional instability, depression and anxiety, changes in sexual desire, physical fatigue, insomnia, and loss of appetite. Behavioral changes are characterized by inattention, accidents, criminality, and suicidal tendencies, and these symptoms disappear after menstruation. The diagnostic basis is that if the above physical, mental and behavioral changes occur repeatedly and periodically during the luteal phase and last for more than three menstrual cycles, premenstrual syndrome can be diagnosed.
Sampling Method: Non-Probability Sample
Enrollment: 266 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
The change of premenstrual syndrome | 4 months
  The Daily Record of Symptom Severity (DRSP) is a tool for assessing symptoms of premenstrual syndrome. The scale contained 14 items, including depression, anxiety and tension, emotional instability, irritability, reduced interest, inattention, lethargy and fatigue, abnormal appetite, abnormal sleep, feeling out of control, body pain and swelling. Each item was scored from 1 to 6 points according to the severity of symptoms (1 = none, 2 = very mild, 3 = mild, 4 = moderate, 5 = severe, 6 = extremely severe). The total score of premenstrual symptoms, physical/emotional/behavioral symptoms and individual index scores were calculated. In this study, participants were asked to fill in the form of the most severe feeling on the 5th day before the menstrual cycle and the previous menstrual cycle before the initiation of the medication at 20:00 to 22:00 every day on the 5th to 9th day of the menstrual cycle to evaluate the changes in symptoms before and after the treatment.

SECONDARY OUTCOMES:
Change of single index of DRSP scale | 4 months
  In DRSP, the scores of premenstrual somatic symptoms, emotional symptoms, and behavioral symptoms, and the scores of individual indicators and their disappearance rates.
Change of TCM premenstrual syndrome | 4 months
  The TCM premenstrual syndrome score scale was designed according to the theory of TCM, which was used to evaluate the TCM syndromes of patients with premenstrual syndrome, including breast swelling and pain, small abdominal distension, irritability, dizziness, insomnia, headache, difficulty in menstruation and other TCM symptoms and signs such as tongue and pulse. The changes of symptom scores of premenstrual syndrome reflect the improvement or deterioration of the condition. The scale uses a semi-quantitative grading method to score the severity of different symptoms into 0, 2, 4, and 6 points (such as breast pain, etc.) or 0, 1, 2, and 3 points (such as dizziness, etc.). The lowest score was 0, and the highest specific score was determined according to the accumulation of each symptom score. The higher the score, the more severe the condition. The reduction rate of TCM syndrome and the disappearance rate of single symptom in the TCM syndrome score table were calculated.

IPD SHARING:
Plan to Share IPD: No